CLINICAL TRIAL: NCT02951416
Title: The European IPF Registry - an Internet-based, Pan-European Registry Linked to the European IPF Biobank (eurIPFbank)
Brief Title: Clinical Course of Interstitial Lung Diseases: European IPF Registry and Biobank
Acronym: eurIPFreg
Status: Active, not recruiting | Type: Observational
Sponsor: Andreas Guenther (Other)
Responsible Party: Sponsor-Investigator, Andreas Guenther, Professor of Internal Medicine, University of Giessen
Organization: University of Giessen (Other)
Other Study IDs: EurIPFreg_150609
Record Dates: First submitted 2015-06-09; First posted 2016-11-01 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Idiopathic Pulmonary Fibrosis; Idiopathic Interstitial Pneumonia; Interstitial Lung Diseases; Diffuse Parenchymal Lung Diseases
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Idiopathic Interstitial Pneumonias; Lung Diseases, Interstitial | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Biospecimen Retention: Samples With DNA — EDTA blood, Plasma, Serum, GenePAX blood, BALF, BALCP, lung tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (15):
- Idiopathic Pulmonary Fibrosis (IPF): IPF diagnosis according to the guidelines of 2011 (AJRCCM 2011; 183:788). For patients diagnosed prior to 2011, the criteria of the consensus statement 2000 apply (AJRCCM 2000;161:646).
  Patient registry (observation and biomaterial sampling).
  Interventions: Other: patient registry (observation and biomaterial sampling)
- Non-specific interstitial pneumonia: Non-specific interstitial pneumonia (NSIP) based on the histopathological demonstration of an NSIP pattern.
  Patient registry (observation and biomaterial sampling).
  Interventions: Other: patient registry (observation and biomaterial sampling)
- Cryptogenic organising pneumonia (COP): COP characterised histologically by an organising pneumonia with intraluminal organising fibrosis in the alveolar ducts and alveolar spaces.
  Patient registry (observation and biomaterial sampling).
  Interventions: Other: patient registry (observation and biomaterial sampling)
- Acute interstitial pneumonia (AIP): Histological pattern of diffuse alveolar damage (DAD), characterised by hyaline membranes, alveolar oedema and a marked interstitial and alveolar inflammatory reaction.
  Patient registry (observation and biomaterial sampling).
  Interventions: Other: patient registry (observation and biomaterial sampling)
- Lymphoid interstitial pneumonia (LIP): Histological pattern of LIP primary or secondary (e.g. rheumatoid arthritis, Sjögren's syndrome, pernicious anaemia, chronic active hepatitis, systemic lupus erythematosus (SLE), primary biliary cirrhosis, myasthenia gravis, severe immune deficiency syndromes (AIDS)).
  Patient registry (observation and biomaterial sampling).
  Interventions: Other: patient registry (observation and biomaterial sampling)
- respiratory bronchiolitis-ILD (RB-ILD): Histological pattern of RB-ILD or typical clinical and radiological findings. Patient registry (observation and biomaterial sampling).
  Interventions: Other: patient registry (observation and biomaterial sampling)
- Desquamative Interstitial Pneumonia: Histological pattern of Desquamative Interstitial Pneumonia (DIP). The picture is similar to RB-ILD, but the distribution pattern is much more homogeneous and does not even have the bronchiolocentric distribution.
  Patient registry (observation and biomaterial sampling).
  Interventions: Other: patient registry (observation and biomaterial sampling)
- Hypersensitivity Pneumonitis: Hypersensitivity Pneumonitis (HP) characterized by exposure to inhaled organic antigens and development of antibodies. Typical clinical and radiological findings, lymphocytosis in bronchoalveolar lavage (BAL) or histology showing HP granulomas.
  Patient registry (observation and biomaterial sampling).
  Interventions: Other: patient registry (observation and biomaterial sampling)
- Sarcoidosis: Histological pattern with sarcoid granulomas or typical clinical and radiological findings with a lymphocytosis in BAL.
  Patient registry (observation and biomaterial sampling).
  Interventions: Other: patient registry (observation and biomaterial sampling)
- Lung Cancer: Histological confirmation of Lung Cancer. Patients will be included as control group.
  Patient registry (observation and biomaterial sampling).
  Interventions: Other: patient registry (observation and biomaterial sampling)
- Chronic Obstructive Pulmonary Disease: Obstructive spirometry and physical history suggesting Chronic Obstructive Pulmonary Disease (COPD). Patients will be included as control group.
  Patient registry (observation and biomaterial sampling).
  Interventions: Other: patient registry (observation and biomaterial sampling)
- Pulmonary Hypertension: Pulmonary Hypertension (PH) diagnosed through right heart catheterisation. Patients will be included as control group.
  Patient registry (observation and biomaterial sampling).
  Interventions: Other: patient registry (observation and biomaterial sampling)
- Sleep Apnea: Sleep Apnea diagnosed by polysomnography. Patients will be included as control group.
  Patient registry (observation and biomaterial sampling).
  Interventions: Other: patient registry (observation and biomaterial sampling)
- Asthma: Asthma diagnosed by positive bronchoprovocation test and typical history or bronchoreversibility in the lung function measurement or through peak flow measurement. Patients will be included as control group.
  Patient registry (observation and biomaterial sampling).
  Interventions: Other: patient registry (observation and biomaterial sampling)
- Control/Health Individuals: Healthy volunteers not suffering from any lung disease as control group. Patient registry (observation and biomaterial sampling).
  Interventions: Other: patient registry (observation and biomaterial sampling)

INTERVENTIONS:
Other: patient registry (observation and biomaterial sampling) — data are collected with patient questionnaires, additionally clinical data are collected at every routine visit and biomaterial is collected

SUMMARY:
Born out of the European Union 7th Framework Programme funded project European IPF Network (eurIPFnet), the European IPF Registry (eurIPFreg) has become Europe's leading database of longitudinal data from IPF patients, including control groups of patients with other lung diseases. The registry was initiated with the intention of creating a permanent and continuously growing record of well defined data on IPF in Europe, in order to increase the chances of finding better treatment options for this devastating disease.

Clinical colleagues who would like to actively participate (both in terms of patient recruitment and data analysis) are invited to contact us (http://www.pulmonary-fibrosis.net/).

DETAILED DESCRIPTION:
The group's work aims to foster research on Idiopathic Pulmonary Fibrosis (IPF), the most aggressive form of an Idiopathic Interstitial Pneumonia (IIP). Within the eurIPFreg we, the eurIPFreg steering committee and a growing number of external site investigators, aim to describe the natural course of IPF and other IIPs, to identify risk factors that are associated with the evolution of the disease and to sample biomaterials that may serve as underlying basis for translational research activities.

IPF and non-specific interstitial pneumonia (NSIP), as well as the other entities of IIPs (cryptogenic organizing pneumonia, COP; desquamative interstitial pneumonia, DIP; respiratory bronchiolitis interstitial lung disease, RB-ILD; lymphoid interstitial pneumonia, LIP; acute interstitial pneumonia, AIP) are frequently progressive, fibroproliferative diseases of unknown etiology, affecting the lung parenchyma. Patients with IPF have the most devastating prognosis within the group of IIPs, with a median survival rate of 2-3 years.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed

Exclusion Criteria:

* No informed consent signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Interstitial Lung Diseases
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2009-09; Primary Completion 2025-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
clinical course of patients with Interstitial Lung Diseases (ILD) | 5 years
  change of lung function parameter such as forced vital capacity (FVC), diffusing lung capacity (DLCO) over time mortality symptoms (reported in patients questionnaires)

SECONDARY OUTCOMES:
Comorbidities of patients with ILD | 5 years
  reported in patients and physicians questionnaires
Infections in lung function of patients with ILD | 5 years
  reported in patients and physicians questionnaires
Quality of life of patients with ILD | 5 years
  reported in patients and physicians questionnaires, EQ5D (European quality of life 5-dimensions) questionnaire
Health care utilization of patients with ILD | 5 years
  reported in patients questionnaires

CONTACTS AND LOCATIONS:
Locations (7):
- Medizinische Universität Wien, Vienna, Austria
- France (2):
  - Centre Hospitalier Universitaire Dijon, Dijon
  - Hopital Bichat Paris, Paris
- Germany (2):
  - Andreas Guenther, Giessen
  - Lungenfachklinik Waldhof Elgershausen, Greifenstein
- Università degli Studi di Catania, Catania, Italy
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guenther A; European IPF Network. The European IPF Network: towards better care for a dreadful disease. Eur Respir J. 2011 Apr;37(4):747-8. doi: 10.1183/09031936.00012111. No abstract available. PMID 21454892
- [Background] Loeh B, Drakopanagiotakis F, Bandelli GP, von der Beck D, Tello S, Cordani E, Rizza E, Barrocu L, Markart P, Seeger W, Guenther A, Albera C. Intraindividual response to treatment with pirfenidone in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2015 Jan 1;191(1):110-3. doi: 10.1164/rccm.201406-1106LE. No abstract available. PMID 25551350
- [Derived] Krauss E, Claas LH, Tello S, Naumann J, Wobisch S, Kuhn S, Majeed RW, Moor K, Molina-Molina M, Byrne O, Borton R, Wijsenbeek MS, Hirani N, Vancheri C, Crestani B, Guenther A; eurILDreg investigators. European ILD registry algorithm for self-assessment in interstitial lung diseases (eurILDreg ASA-ILD). PLoS One. 2025 Jan 29;20(1):e0316484. doi: 10.1371/journal.pone.0316484. eCollection 2025. PMID 39879227
- [Derived] Krauss E, Tello S, Naumann J, Wobisch S, Ruppert C, Kuhn S, Mahavadi P, Majeed RW, Bonniaud P, Molina-Molina M, Wells A, Hirani N, Vancheri C, Walsh S, Griese M, Crestani B, Guenther A; further eurILDreg investigators; RARE-ILD investigators. Protocol and research program of the European registry and biobank for interstitial lung diseases (eurILDreg). BMC Pulm Med. 2024 Nov 18;24(1):572. doi: 10.1186/s12890-024-03389-9. PMID 39558302
- [Derived] Krauss E, Haberer J, Barreto G, Degen M, Seeger W, Guenther A. Recognition of breathprints of lung cancer and chronic obstructive pulmonary disease using the Aeonose(R) electronic nose. J Breath Res. 2020 Jul 24;14(4):046004. doi: 10.1088/1752-7163/ab8c50. PMID 32325432
- [Derived] Krauss E, Gehrken G, Drakopanagiotakis F, Tello S, Dartsch RC, Maurer O, Windhorst A, von der Beck D, Griese M, Seeger W, Guenther A. Clinical characteristics of patients with familial idiopathic pulmonary fibrosis (f-IPF). BMC Pulm Med. 2019 Jul 18;19(1):130. doi: 10.1186/s12890-019-0895-6. PMID 31319833
- [Derived] Witt S, Krauss E, Barbero MAN, Muller V, Bonniaud P, Vancheri C, Wells AU, Vasakova M, Pesci A, Klepetko W, Seeger W, Crestani B, Leidl R, Holle R, Schwarzkopf L, Guenther A. Psychometric properties and minimal important differences of SF-36 in Idiopathic Pulmonary Fibrosis. Respir Res. 2019 Mar 1;20(1):47. doi: 10.1186/s12931-019-1010-5. PMID 30823880
- [Derived] Loeh B, Brylski LT, von der Beck D, Seeger W, Krauss E, Bonniaud P, Crestani B, Vancheri C, Wells AU, Markart P, Breithecker A, Guenther A. Lung CT Densitometry in Idiopathic Pulmonary Fibrosis for the Prediction of Natural Course, Severity, and Mortality. Chest. 2019 May;155(5):972-981. doi: 10.1016/j.chest.2019.01.019. Epub 2019 Feb 8. PMID 30742809
- [Derived] Guenther A, Krauss E, Tello S, Wagner J, Paul B, Kuhn S, Maurer O, Heinemann S, Costabel U, Barbero MAN, Muller V, Bonniaud P, Vancheri C, Wells A, Vasakova M, Pesci A, Sofia M, Klepetko W, Seeger W, Drakopanagiotakis F, Crestani B. The European IPF registry (eurIPFreg): baseline characteristics and survival of patients with idiopathic pulmonary fibrosis. Respir Res. 2018 Jul 28;19(1):141. doi: 10.1186/s12931-018-0845-5. PMID 30055613
- See also: European IPF Registry website — http://www.pulmonary-fibrosis.net/